CLINICAL TRIAL: NCT06624865
Title: Microbiota and Carcinogenesis of Small-intestine Neuroendocrine Tumors
Acronym: Microbio-siNET
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1290; 2023-A02667-38 (Other: ANSM)
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Small-intestine Neuroendocrine Tumors
Keywords: Small-intestine neuroendocrine tumor; microbiota; tumorigenesis
MeSH Terms: conditions — Carcinogenesis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Blood and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient with indication for small-intestine neuroendocrine tumor surgery: The target population for this study is consecutive patients with small-intestine neuroendocrine tumor for whom surgery is indicated
  Interventions: Other: Blood and stool sampling

INTERVENTIONS:
Other: Blood and stool sampling — Blood and stool sampling

SUMMARY:
The aim of the study is to investigate the impact of the microenvironment on tumorigenesis of small intestinal neuroendocrine tumors often located in the terminal ileum, without identified driver mutations.

ELIGIBILITY:
Inclusion Criteria:

* Patient with one or more small-intestine neuroendocrine tumor with indication of surgery
* Patient with consent for the collection, storage and reuse of data associated with his/her disease
* Age ≥ 18 years at the time of inclusion
* Non-objection statement obtained for participation in the study

Exclusion Criteria:

* Patients with poorly differentiated neuroendocrine carcinoma or NET (neuroendocrine tumors) of non-intestinal origin or mixed tumors (MiNEN)
* Pregnant, parturient or breast-feeding women
* Minors
* Persons deprived of liberty by judicial or administrative decision
* Adults under legal protection (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients followed at the Edouard Herriot University Hospital with small-intestine neuroendocrine tumors of the small intestine and indication for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Composition of microbiota | At day 1 and month 3
  Determination of the composition of blood, fecal, intra- and peri-tumoral microbiota in patients undergoing surgery for small-intestine neuroendocrine tumor.

CONTACTS AND LOCATIONS:
Locations (1):
- Edouard Herriot University Hospital, Lyon, France, France